CLINICAL TRIAL: NCT07182253
Title: Effects of Ashwagandha Extract (Capsule KSM-66 300 mg) on Sexual Health in Healthy Women: A Prospective, Randomized, Double-Blind, Placebo- Controlled Study
Brief Title: Effect of Single Dose of Ashwagandha Root Extract on Sexual Health in Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ixoreal-FSD-CT-1022
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Female Sexual Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1: Interventional KSM-66 Ashwagandha® capsule (300 mg) (Active Comparator): KSM-66 Ashwagandha root extract
  Interventions: Dietary Supplement: KSM-66 Ashwagandha® capsule
- Treatment Arm 2: Identical placebo capsule (Placebo Comparator): Starch
  Interventions: Other: Identical Placebo capsule

INTERVENTIONS:
Dietary Supplement: KSM-66 Ashwagandha® capsule — Two off-white capsules, each containing 300 mg KSM-66 Ashwagandha root extract powder only.
  Arms: Treatment Arm 1: Interventional KSM-66 Ashwagandha® capsule (300 mg)
Other: Identical Placebo capsule — Two off-white capsules containing starch powder only
  Arms: Treatment Arm 2: Identical placebo capsule

SUMMARY:
Sexual health is a key part of a woman's overall physical, emotional, and mental well-being-even in the absence of any medical or psychological problems. It includes aspects such as sexual desire, arousal, satisfaction, and confidence in intimate relationships. Everyday factors like stress, fatigue, work-life balance, and hormonal changes can impact these areas, even in otherwise healthy women. Unfortunately, sexual wellness is often under-discussed in both clinical practice and research, especially for women who are not experiencing a diagnosed disorder.

This study is designed to explore whether Ashwagandha root extract (KSM-66), a natural herbal supplement known for its stress-reducing and vitality-enhancing properties, can help support and maintain sexual wellness in healthy adult women. Unlike treatments aimed at correcting dysfunction, this research focuses on enhancing natural sexual function-improving desire, mood, and satisfaction as part of overall health. Participants take either Ashwagandha or a placebo over several weeks, and their experiences are measured using validated tools like the Female Sexual Function Index (FSFI).

Understanding and supporting sexual wellness through natural means can improve not only intimacy and relationship satisfaction, but also self-esteem, mood, and general life satisfaction. By addressing sexual health proactively in healthy individuals, this study contributes to a more complete picture of women's health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female participants between 18 to 55 years of age. 2. The participate should inform their partner about the study 3. Her partner should be willing to let her participate in the study 4. Participants willing to try to have sexual intercourse regularly. 5. Participants in a stable, monogamous, heterosexual relationship that is secure and communicative, for at least 6 months prior to the Screening Visit.

  6. Participant's partner is expected to be physically present at least 50% of each month.

  7. Participants who have used a medically acceptable method of contraception for at least 3 months before the baseline Visit (Visit 1) and continue to use that medically acceptable method of contraception during the trial.

  8. Participants who are reliable, honest, compliant, and agree to co-operate with all trial evaluations as well as to be able to perform them as per investigator's opinion.

  9. Participants or LAR can and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements.

  10. Participants having sufficient understanding to communicate effectively with the investigator and are willing to discuss their sexual functioning with the investigative staff.

  11. Participants who are willing to have 4 or more attempts of sexual intercourse each month.

Exclusion Criteria:

* 1. Participants who are not willing to take an investigational product. 2. Any acute illness which may hamper the study participation as per principal investigator discretion at the time of enrolment.

  3. Participants having any clinically significant medical history, medical finding or an on- going medical or psychiatric condition exists which in the opinion of the Investigator could jeopardize the safety of the subject, impact validity of the study results or interfere with the completion of study according to the protocol.

  4. Individuals participating in any other studies, including macro/micro/any other forms of dietary supplements/multivitamins or disease-specific oral nutrition supplements (for improving the sexual function during the 3 months prior to study commencement).

  5. Participants having a history of hypersensitivity reactions (i.e., allergic or oversensitivity to usual doses).

  6. Participants with current alcohol or drug addiction or with a history of drug dependence or abuse within the past one year.

  7. Participants who indicate that their sexual partner has inadequately treated sexual problems that could interfere with the Subjects response to treatment.

  8. Participants who have entered the menopausal transition or menopause or have had a hysterectomy.

  9. Participants with findings of infection, inflammation, undue tenderness, or shrinkage (atrophy) of the female genital organs, at the Screening Visit.

  10. Participants who are breastfeeding or have breastfed within the last 6 months prior to the Baseline Visit.

  11. Participants who are pregnant or have been pregnant within the last 6 months prior to the Baseline Visit.

  12. Participants having primary hypoactive sexual desire. 13. Participants with a history of malignancy. 14. Participate itself are not planning to get pregnant for next six months 15. Participants who cannot cooperate to complete the subject records during the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of the KSM-66 Ashwagandha formulation on sexual health in healthy women, assessed based on Female Sexual Function Index (FSFI) in healthy women | Baseline, Week 4, Week 8
  Mean change in FSFI scores from Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4) to Visit 3- End of study (Week 8) in healthy women

SECONDARY OUTCOMES:
To evaluate the effects of the KSM-66 Ashwagandha formulation on sexual health in healthy women, assessed based on the Satisfying Sexual Events (SSEs) in healthy women | Baseline, Week 4, Week 8
  Mean change in SSEs from Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4) to Visit 3- End of study (Week 8) in healthy women
To evaluate the effects of the KSM-66 Ashwagandha formulation on sexual health in healthy women, assessed based on the Female Sexual Distress Scale (FSDS) in healthy women | Baseline, Week 4, Week 8
  Mean change in FSDS scores from Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4) to Visit 3- End of study (Week 8) in healthy women
To investigate the effects of KSM-66 Ashwagandha formulation on serum hormones (Estrogen-E2, Progesterone, FSH, LH, Prolactin, and Testosterone) in healthy women | Baseline, Week 4, Week 8
  Mean change in serum hormones (Estrogen-E2, Progesterone, FSH, LH, Prolactin, and Testosterone) from Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1) to Visit 3- End of study (Week 8) in healthy women
To evaluate the effects of KSM-66 Ashwagandha formulation on stress using the Perceived Stress Scale (PSS-10) | Baseline, Week 4, Week 8
  Mean change in PSS-10 scores from Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4) to Visit 3- End of study (Week 8) in healthy women
To evaluate the effect of the KSM-66 Ashwagandha formulation on Quality of Life (SF-12 QoL) in healthy women | Baseline, Week 4, Week 8
  Mean change in SF-12 scores from Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4) to Visit 3- End of study (Week 8) in healthy women
To evaluate the safety of KSM-66 Ashwagandha formulation in healthy women | Baseline, Week 4, Week 8
  Number and proportion of Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Event (TESAE) over 8 weeks treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States